CLINICAL TRIAL: NCT01961050
Title: Preventing FAS/ARND in Russian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Fogarty International Center of the National Institute of Health (NIH); St. Petersburg State Pavlov Medical University (Other); Nizhny Novgorod State Pedagogical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AA016234_IRB 2758; 5R01AA016234 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Fetal Alcohol Syndrome (FAS); Fetal Alcohol Spectrum Disorders; Alcohol Abuse in Pregnancy
Keywords: alcohol; pregnancy; fetal exposure; prevention; FAS; Alcohol-Related Neurodevelopmental Disorder (ARND)
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Dual-Focused Brief Physician Intervention (DFBPI)
  Interventions: Behavioral: Dual-Focused Brief Physician Intervention (DFBPI)
- Standard care (Other): Services as usual including standard OB/GYN clinic visits; no experimental intervention is provided.
  Interventions: Other: Services as usual

INTERVENTIONS:
Behavioral: Dual-Focused Brief Physician Intervention (DFBPI) — The DFBPI is incorporated in OB/GYN clinic visit. The intervention consists of two brief (5 to 10 minutes) manualized counseling segments delivered face-to-face by an OB/GYN in the context of two clinic visits.
  Arms: Intervention
Other: Services as usual — Active Comparator: Standard OB/GYN clinic visits that include OB/GYN services as usual.
  Arms: Standard care

SUMMARY:
The purpose of this study is to evaluate an intervention aimed at reducing risk for alcohol-exposed pregnancies and preventing Fetal Alcohol Spectrum Disorders in Russian children. The study will determine whether physicians, trained in a dual-focused brief motivational intervention and monitored for performance, can foster greater change in knowledge, health beliefs, alcohol use, and alcohol-exposed pregnancy risk in Russian women who are at risk than standard care.

DETAILED DESCRIPTION:
The study is a two-arm, 20-site, site-randomized, controlled trial testing an intervention to reduce risk for alcohol-exposed pregnancies in at-risk women (at-risk drinking childbearing age women who are heterosexually active, and not consistently using contraception). The trial will assess feasibility of a dual-focused (i.e. contraception use-drinking reduction) brief physician intervention (DFBPI) and determine whether physicians, trained in DFBPI and monitored for compliance, can foster greater reduction of women's risk behaviors compared to standard care. The intervention is specifically designed to be deliverable routinely by Obstetrics and Gynecology physicians(OB/GYN) to large numbers of women at women's clinics.

ELIGIBILITY:
Inclusion Criteria:

* nonpregnant women
* childbearing age (between 18 and 44 years of age)
* fertile
* at risk for an alcohol-exposed pregnancy: drinking at-risk (4 or more drinks on one occasion or more than 7 drinks per week)in the last 3 months and report having unprotected intercourse at least once in the last 6 months

Exclusion Criteria:

* unable comprehend interview questions

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 767 (Actual)
Dates: Start 2007-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Alcohol-Exposed Pregnancy (AEP) risk at 3 months | 3 months
  Interviews are conducted at the baseline and follow-up assessments at 3, 6, and 12 months after the baseline to assess self-reported alcohol consumption, sexual activity, and contraception use to identify AEP risk.
Change from Baseline Alcohol-Exposed Pregnancy (AEP) risk at 6 months | 6 months
  Interviews are conducted at the baseline and follow-up assessments at 3, 6, and 12 months after the baseline to assess self-reported alcohol consumption, sexual activity, and contraception use to identify AEP risk.
Change from Baseline Alcohol-Exposed Pregnancy (AEP) risk at 12 months | 12 months
  Interviews are conducted at the baseline and follow-up assessments at 3, 6, and 12 months after the baseline to assess self-reported alcohol consumption, sexual activity, and contraception use to identify AEP risk.

SECONDARY OUTCOMES:
Changes in alcohol consumption from baseline | 3 months, 6 months, and 12 months follow-up
  Interviews assessed self-reported quantity/frequency of alcohol consumption and frequency of binge drinking and a detailed alcohol consumption report was received utilizing the Time Line Follow Back (TLFB) measure.
Changes in knowledge about Fetal Alcohol Syndrome (FAS) from baseline | 3 months, 6 months, and 12 months follow-up
  A survey measure assessed knowledge about FAS
Changes in Health beliefs and attitudes from baseline | 3 months, 6 months, and 12 months follow-up
  A survey measure assessed attitudes and health beliefs related to alcohol use during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Balachova, PhD, Principal Investigator — University of Oklahoma
Locations (2):
- Russia (2):
  - Women's Clinics, Nizhny Novgorod
  - Women's clinics, Saint Peterburg

REFERENCES:
- [Result] Balachova T, Bonner BL, Chaffin M, Isurina G, Shapkaitz V, Tsvetkova L, Volkova E, Grandilevskaya I, Skitnevskaya L, Knowlton N. Brief FASD prevention intervention: physicians' skills demonstrated in a clinical trial in Russia. Addict Sci Clin Pract. 2013 Jan 8;8(1):1. doi: 10.1186/1940-0640-8-1. PMID 23294846